CLINICAL TRIAL: NCT02843646
Title: Investigating the Use of the WalkAide on a Child's Ability to Ascend/Descend Stairs and Curbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blythedale Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Walk_Aide
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
Keywords: gait training; stepping
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walk Aide training (Experimental): This group of children will receive six weeks of Walk Aide training. During training, children will wear the Walk Aide. This device triggers ankle dorsiflexion, and controls the timing and duration of personal nerve stimulation during the swing phase of gait. The duration of the stimulus is gradually increased along with the wearing of the Walkaide. Subjects will begin by wearing the prosthesis for 30 minutes. The wearing time will be increased to waking hours of the subject, depending on their age. The electrodes will be placed on the client before the session is to begin, and taken off immediately after WalkAide usage. The skin will be checked before and after WalkAide electrode usage. The skin will be cleaned with an alcohol wipe before the electrodes are applied.
  Interventions: Device: Walk Aide training
- Delayed Walk Aide training (Placebo Comparator): This group of children will not receive Walk Aide training during the first six weeks of enrollment. This group will serve as a comparator group to Arm 1. After six weeks, children in this group will be given the option to complete the 6-week Walk Aide training protocol that is given in Arm 1.
  Interventions: Device: Walk Aide training

INTERVENTIONS:
Device: Walk Aide training

SUMMARY:
The purpose of this study is to investigate the use of the WalkAide, a Neuroprosthetic device, on a child's ability to ascend/descend stairs and curbs. It is hypothesized that with WalkAide use, the improved ankle control achieved, will affect the speed, symmetry, and independence of completing the task.

DETAILED DESCRIPTION:
The investigators will examine the use of the WalkAide, a Neuroprosthetic device, on a child's ability to ascend/descend stairs and curbs. It is hypothesized that with WalkAide use, the improved ankle control achieved, will affect the speed, symmetry, and independence of completing the task.

Study subjects will be fitted with the WalkAide by Physical Therapists trained in this procedure. Subjects will build tolerance to the device over a two-week period, and use as able for the next six weeks. The children (participants/subjects) in the study will go through a desensitization process to familiarize them with the electrical stimulation.

The children will begin with no stimulation, wearing the Walkaide to introduce the sensation of the cuff on their leg prior to beginning the stimulation. Once familiar with the feel of the Walkaide, the electrical stimulation will be introduced slowly and gradually. The child's face and verbal responses will be monitored while the stimulation is introduced and turned up to the desired response threshold.

An age and cognitively appropriate pain scale will be available if applicable to the child and situation.

The children will be assured that if they do not want to continue or if they feel uncomfortable, then the electrical stimulation will be turned off immediately. The minimum stimulus intensity is determined in collaboration with each subject. The children are asked to identify when they first begin to feel the stimulus, and the number on the intensity knob is noted. The duration of the stimulus is gradually increased along with the wearing of the Walkaide. Subjects will begin by wearing the prosthesis for 30 minutes. The wearing time will be increased to waking hours of the subject, depending on their age. The electrodes will be placed on the client before the session is to begin, and taken off immediately after WalkAide usage. The skin will be checked before and after WalkAide electrode usage. The skin will be cleaned with an alcohol wipe before the electrodes are applied. It is normal to observe somewhat reddened areas under the electrode placement following usage. However, the redness should disappear within an hour. With signs of irradiation or maintained redness, small pimple like lesions or blisters, the WalkAide usage will be discontinued at that time, and the patient will be brought to the medical staff. The skin will be re-evaluated an hour later following the electrode usage. The Pediatrician for that patient will be immediately notified, and the WalkAide usage discontinued until the problem is resolved.

ELIGIBILITY:
Inclusion Criteria:

* Ability to ambulate independently with or without an assistive device and/or lower extremity orthoses.
* Ability to follow and understand experimental procedures.

Exclusion Criteria:

* Seizure history interfering with use of functional electrical stimulation as verified by their MD.
* Inability to be able to complete the assessment tests to gain a baseline score.
* Skin irritation/skin intact.
* Uncorrected vision impairments.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2016-07; Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in the Timed-Up-and-Down-Stairs (TUDS) measure | Day 1 of intervention and up to 5 days after the last day of intervention
  Measures the ability of a child to negotiate stairs
Change in the Step-Up-and-Over measure | Day 1 of intervention up to 5 days after the last day of intervention
  Measures the ability of a child to step up and over a curb

SECONDARY OUTCOMES:
Pain scale | Each day of therapy, from date of randomization until up to six weeks after date of randomization
  Children will be asked to rate pain caused by the Walk Aide on each day of therapy (day of therapy only)

CONTACTS AND LOCATIONS:
Locations (1):
- Blythedale Children's Hospital, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided